CLINICAL TRIAL: NCT05721716
Title: A Feasibility Randomised Controlled Trial of a Mindfulness Booster Course Following an 8-week Staff Mindfulness Programme
Brief Title: Examining the Feasibility of a Mindfulness Booster Course for Healthcare Staff Who Attended an 8-week Mindfulness Course
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canterbury Christ Church University (Other)
Collaborators: Sussex Partnership NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DClinPsychol21KWalker
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Stress

STUDY DESIGN:
Masking Description: Assessment of outcome will be by self-report measures administered by an online survey. Therefore, assessment of outcome will be masked from the researchers, but not the participants themselves.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Booster Course (Experimental)
  Interventions: Behavioral: Mindfulness Booster Course; Behavioral: Usual care
- Treatment as Usual Control (Other)
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Mindfulness Booster Course — The mindfulness booster course will consist of eight 30-minute sessions, which participants will be asked to commit to. These will be online and occur weekly for 8-weeks. Within these sessions, there will be a 15-minute mindfulness practice followed by a 15-minute discussion. This discussion time will involve reflecting on the mindfulness practice and speaking about between-session practice. Participants will be encouraged to practice mindfulness for home work between the sessions.
  Arms: Mindfulness Booster Course
Behavioral: Usual care — Participants will be encouraged to continue with whatever activities they usually undertake to manage their stress and support their wellbeing.

SUMMARY:
The goal of this clinical trial is to examine the feasibility and acceptability of a mindfulness booster course for UK healthcare staff who have previously participated in an eight-week mindfulness course. The measures of feasibility and acceptability that will be examined include: 1. the ease with which participants are recruited to the clinical trial; 2. the extent to which participants choose to remain in the mindfulness booster course; 3. the extent to which participants choose to remain in the clinical trial; 4. how acceptable the participants find the mindfulness booster course; 5. the level of outcome measure completion; 6. whether there is a preliminary indication that the course may reduce stress. Participants will be randomly allocated to either a mindfulness booster course or a control group, who will be encouraged to continue taking care of their wellbeing as they normally would. Participants will be asked to complete questionnaires at three time-points.

DETAILED DESCRIPTION:
This pilot randomised controlled trial seeks to examine the feasibility and acceptability of a mindfulness booster course for UK National Health Service staff who have previously completed an 8-week mindfulness-based intervention. Participants will be randomised to either the 8-week mindfulness booster course or a control group, in which participants will be encouraged to continue taking care of their wellbeing as they normally would. A battery of self-report measures will be administered online at baseline (weeks 0-1), mid-intervention (week 7), and post-intervention (weeks 11-12). The indices of feasibility and acceptability that will be examined include: 1. ease of recruitment; 2. participant retention in the intervention; 3. participant retention in the study; 4. acceptability of the intervention; 5. outcome measure completion; 6. whether there is a preliminary signal of efficacy on the primary outcome measure (stress). These indices will be compared to progression criteria (which are detailed in the outcome measures section) to determine whether the intervention is sufficiently feasible and acceptable to progress to a full-scale RCT in future research.

ELIGIBILITY:
Inclusion Criteria:

* UK National Health Service staff member from the South-East, South-West and/or London, including, but not limited to, Sussex Partnership NHS Foundation Trust;
* have completed an 8-week staff mindfulness course within the past three-years (individuals will be considered to have "completed" a mindfulness course if they attended four or more sessions (Simpson et al., 2017; Verweij et al., 2018)).

Exclusion Criteria:

* currently on sick leave;
* planning on undertaking another 8-week mindfulness course;
* have previously found practicing mindfulness distressing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited | 10 months following the start of recruitment
  The number of participants recruited over 10-months will be compared against the following progression criterion to assess the feasibility of recruitment: Green: 40-50; Amber 24-39; Red: <24.
Proportion of intervention group participants who attend at least half of the mindfulness booster course intervention sessions | Weeks 0 to 12
  The proportion of participants who attend at least half of the intervention sessions will be compared against the following progression criterion to assess retention in the intervention: Green: ≥50%; Amber 25-49%; Red: <25%.
Proportion of study participants who remain in the study | Weeks 0 to 12
  The proportion of study participants who remain in the study will be compared against the following progression criterion to assess retention in the study: Green: ≥50%; Amber 25-49%; Red: <25%.
Mindfulness booster course acceptability | Weeks 11 to 12
  Response to Likert type questions and content analysis of qualitative data will be compared against the following progression criterion to assess retention in the study: Green: the majority of intervention participants report the intervention is acceptable as it is or with minor adjustments; Amber: there are inconsistent reports of acceptability or the intervention requires bigger adjustments; Red: the majority of intervention participants report the intervention is unacceptable or requires adjustments which cannot be completed
Completion rate of the outcome measures | Weeks 0 to 12
  The rate of the outcome measures completion will be compared against the following progression criterion to assess the feasibility of outcome measurement: Green: ≥60%; Amber 40-59%; Red: <40%.
Estimate of between group effect size of the mindfulness booster intervention compared to control on the primary outcome measure of change in Perceived Stress Scale scores from baseline (weeks 0-1) to post-intervention (weeks 11-12). | Weeks 11-12
  The estimated between group effect size of the mindfulness booster intervention compared to control on the primary outcome measure of change in Perceived Stress Scale scores from baseline (weeks 0-1) to post-intervention (weeks 11-12) will be compared against the following progression criterion to provide a preliminary indicator of effectiveness: Green: effect size in favour of intervention arm and 95% confidence interval for that effect size contains (or is greater than) the minimal clinically important difference found by Drachev et al. (2020). Amber: effect size is in favour of control, but the minimum clinically important difference is included in the 95% confidence interval; Red: effect size is in favour of control, and the minimum clinically important difference is not included in the 95% confidence interval.

SECONDARY OUTCOMES:
Estimate of the between group effect size of the mindfulness booster intervention compared to control on change in the 8-item Patient Health Questionnaire (PHQ-8) from baseline (weeks 0-1) to post-intervention (weeks 11-12). | Weeks 11-12
  The 8-item Patient Health Questionnaire (PHQ-8) is a self-report measure of depression, with higher scores indicating greater levels of depression symptoms.
Estimate of the between group effect size of the mindfulness booster intervention compared to control on change in the 7-item Generalised Anxiety Disorder Scale (GAD-7) from baseline (weeks 0-1) to post-intervention (weeks 11-12). | Weeks 11-12
  The 7-item Generalised Anxiety Disorder Scale (GAD-7) is a self-report measure of generalised anxiety, with higher scores indicating greater levels of generalized anxiety symptoms.
Estimate of the between group effect size of the mindfulness booster intervention compared to control on change in the 15-item Five-Facet Mindfulness Questionnaire (FFMQ-15) from baseline (weeks 0-1) to post-intervention (weeks 11-12). | Weeks 11-12
  The 15-item Five-Facet Mindfulness Questionnaire (FFMQ-15) is a self-report measure of mindfulness, with higher scores indicating greater levels of mindfulness.
Estimate of the between group effect size of the mindfulness booster intervention compared to control on change in the Brief Sussex Oxford Compassion to Self Scale (SOCS-S) from baseline (weeks 0-1) to post-intervention (weeks 11-12). | Weeks 11-12
  The Brief Sussex Oxford Compassion to Self Scale (SOCS-S) is a self-report measure of self-compassion, with higher scores indicating greater levels of self-compassion.
Estimate of the between group effect size of the mindfulness booster intervention compared to control on change in the Brief Compassion for Others Scale (SOCS-O) from baseline (weeks 0-1) to post-intervention (weeks 11-12). | Weeks 11-12
  The Brief Compassion for Others Scale (SOCS-O) is a self-report measure of compassion for others, with higher scores indicating greater levels of compassion.
Estimate of the between group effect size of the mindfulness booster intervention compared to control on change in the Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWS) from baseline (weeks 0-1) to post-intervention (weeks 11-12). | Weeks 11-12
  The Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWS) is a self-report measure of mental wellbeing, with higher scores indicating greater levels of mental wellbeing.
Estimate of the between group effect size of the mindfulness booster intervention compared to control on change in the Sussex Burnout Scale (SBS) from baseline (weeks 0-1) to post-intervention (weeks 11-12). | Weeks 11-12
  The Sussex Burnout Scale (SBS) is a self-report measure of burnout, with higher scores indicating greater levels of burnout.

CONTACTS AND LOCATIONS:
Overall Officials: Fergal Jones, PhD, Study Chair — Canterbury Christ Church University & Sussex Partnership NHS Foundation Trust; Clara Strauss, DPhil, Study Director — Sussex Partnership NHS Foundation Trust & University of Sussex
Locations (1):
- Sussex Mindfulness Centre, Hove, East Sussex, United Kingdom